CLINICAL TRIAL: NCT04296214
Title: Pharmacoeconomics in the Application of 5-azacitidine in the Treatment of Myelodysplastic Syndromes and Acute Myeloid Leukemia
Status: Withdrawn | Type: Observational
Why Stopped: Poor recruitment
Sponsor: Grupo Cooperativo de Hemopatías Malignas (Other)
Responsible Party: Sponsor
Other Study IDs: HAL 318/2019
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Azacitidine 50 mg/m2 for 10 days each 28 days
  Interventions: Drug: 5-azacitidine
- B: Azacitidine 75 mg/m2 for 7 days each 28 days
  Interventions: Drug: 5-azacitidine

INTERVENTIONS:
Drug: 5-azacitidine — Cycles of 28 days

SUMMARY:
The investigators want to compare the global response rate of patients with myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) after six months of treatment with 5-azacitidine on two different doses. First group of 50 mg/m2 for 10 days each 28 days versus 75 mg/m2 for 7 days on 28 days cycles.

DETAILED DESCRIPTION:
5-Azacitidine it's the standard treatment for patients with MDS and it is widely used for AML in patients that aren't fit for intensive treatment. The standard dose of azacitidine is 75 mg/m2 for 7 días on 28 days cycles. Nevertheless there are studies of pharmacokinetics that have showed there is no difference on plasmatic distribution between 25, 50, 75 or 100 mg/m2 with similar concentration curves. The actual presentation of azacitidine is 100 mg per bottle with less of 24 hours of utility after opened. Looking for optimizations on the use of 5-azacitidine, we have changed the dosing to 50 mg/m2 for 10 days on 28 days cycles with a total dose application of 95% of the traditional regimen with the saving of 5 bottles of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of MDS that require treatment with 5-aza characterized by: i) RAEB-1 defined as the presence of 5%-9% of myeloblasts in bone marrow; ii) RAEB-2 defined as the presence of 10%-19% of myeloblasts in bone marrow or 5%-19% blasts in peripheral blood; iii) IPSS-R very high, high or intermediate
* Confirmed AML with blasts ≥ 20% in bone marrow or peripheral blood and that its not candidate to receive intense chemotherapy at consideration of the physician.
* Performance status of 0, 1 o 2 by the Eastern Cooperative Oncology Group (ECOG).
* Availability to sign an informed consent

Exclusion Criteria:

* Previous treatment for MDS or AML with chemotherapy or another antineoplastics including hypomethylating agents.
* Acute promyelocytic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Confirmed diagnosis of MDS that require treatment with 5-aza characterized by: i) RAEB-1 defined as the presence of 5%-9% of myeloblasts in bone marrow; ii) RAEB-2 defined as the presence of 10%-19% of myeloblasts in bone marrow or 5%-19% blasts in peripheral blood; iii) IPSS-R very high, high or intermediate
  2. Confirmed AML with blasts ≥ 20% in bone marrow or peripheral blood and that its not candidate to receive intense chemotherapy at consideration of the physician.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 6 months
  Global response rate by International Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Cooperativo de Hemopatías Malignas, Huixquilucan, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No